CLINICAL TRIAL: NCT04079543
Title: Randomized Controlled Trial of Liberalized NPO Status to Improve Patient Satisfaction in Patients Undergoing Procedures in the Cardiac Catheterization Lab
Brief Title: NPO and Patient Satisfaction in the Cath Lab
Acronym: FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Derek Atkinson, Cardiac Anesthesiologist, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2019-00261
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Patient Satisfaction; Dehydration; Physiological Effects Secondary to Dehydration
Keywords: Nil per os (NPO); TAVR; arrhythmia ablation
MeSH Terms: conditions — Patient Satisfaction; Dehydration

STUDY DESIGN:
Intervention Model Description: Patients will be randomized (1:1) into one of the two groups: Strict NPO (NPO after midnight) or liberal NPO (clear liquids up to 2 hours prior to procedure).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict NPO (Other): NPO after midnight. No solids or liquids after midnight.
  Interventions: Other: NPO past midnight
- Liberal NPO (Other): No solids after midnight. Clear liquids up to 2 hours prior to surgery.
  Interventions: Other: NPO

INTERVENTIONS:
Other: NPO past midnight — NPO after midnight (solids and liquids), except for a sip of water with medication.
  Arms: Strict NPO
Other: NPO — No solids after midnight. Clear liquids up to 2 hours prior to procedure. Patients can take medications with a sip of water.
  Arms: Liberal NPO

SUMMARY:
The purpose of this randomized, control study is to compare liberal vs strict nil per os (NPO) policies on patients undergoing transcatheter aortic valve replacement (TAVR) or arrhythmia ablation. The primary objective of this study is to determine if allowing clear liquids up to 2 hours prior to elective TAVR or elective arrhythmia ablation procedure improves patient satisfaction.

DETAILED DESCRIPTION:
After informed written consent, patients will be randomized into one of the two groups: Strict NPO (NPO after midnight) or liberal NPO (clear liquids up to 2 hours prior to procedure). All patients, regardless of study arm, will be allowed to take medications with a sip of water. All other peri-operative care will be routine. On the day of the procedure, a patient satisfaction survey will be completed and the procedure will be performed as routine.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* patients planned to undergo trans-catheter aortic valve replacement or arrhythmia ablation at Stony Brook University Hospital
* ability to provide written informed consent

Exclusion Criteria:

* Age less than 18 years
* emergency procedure, dysphasia, nutrition administered via feeding tube (NG, PEG, etc.) or intravenously (total parenteral nutrition), gastroparesis,
* patients not alert and oriented to person, place, and date,
* concurrent surgical procedures on the day of TAVR or arrhythmia ablation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-09 (Estimated); Primary Completion 2020-09-09 (Estimated); Study Completion 2021-09-09 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction: survey | Up to 24 hours
  The primary objective is to determine if allowing clear liquids up to 2 hours prior to elective TAVR or elective arrhythmia ablation procedure improves patient satisfaction. Patient satisfaction will be determined by a patient satisfaction survey given 2 hours (+/- 2 hrs) prior to procedure. This survey will assess: thirst, hunger, headache, nausea, lightheadedness, and anxiety.

SECONDARY OUTCOMES:
Exploratory Analyses | Through the end of hospitalization, usually 2 days.
  An independent analysis of each individual component of the satisfaction survey will be performed. Each variable will be scored on a scale of 0-10. Variables: thirst, hunger, headache, nausea, lightheadedness, anxiety.
  * Renal Function
  * Vasopressor Requirement
  * Post-operative nausea and vomiting
  * Post-operative hospital length of stay

REFERENCES:
- [Derived] Atkinson DJ, Romeiser JL, Almasry IO, Tannous HJ, Parikh PB, Bennett-Guerrero E. Randomized controlled trial of liberal vs. standard fasting instructions in percutaneous cardiac procedures. Perioper Med (Lond). 2023 Aug 8;12(1):44. doi: 10.1186/s13741-023-00333-z. PMID 37553699